CLINICAL TRIAL: NCT04790877
Title: Effect of the Consumption of Alcohol-free Beers With Different Carbohydrates Composition on Postprandial Metabolic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Rocio Mateo-Gallego, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PI19/477
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Healthy Diet; Postprandial Hyperglycemia
Keywords: Carbohydrates; Alcohol-free beer; Maltodextrin; Isomaltulose
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Intervention Model Description: The overall study involved two sub-studies. The first one includes 4 arms and the second one includes 5 arms.
Who Masked: Participant, Investigator
Masking Description: The investigator who prepares the beverages and the bread is not blinded but the investigator who manage the samples and is plan to analyze the results is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- First sub-study: Glucose beverage (Active Comparator): This intervention entails the intake of a beverage including 25 g of glucose.
  Interventions: Other: Sub-study 1
- First sub-study: Regular alcohol-free beer (Experimental): This intervention entails the intake of regular alcohol-free beer including 25 of carbohydrates.
  Interventions: Other: Sub-study 1
- First sub-study: Alcohol-free beer with modified composition (isomaltulose + maltodextrin) (Experimental): This intervention entails the intake of an alcohol-free beer with modified composition in which the maltose has been almost completely eliminated and enriched with isomaltulose (2.5 g/100 mL) and a resistant maltodextrin (0.8 g/100 mL) (IMB). This beverage included 25 g of carbohydrates.
  Interventions: Other: Sub-study 1
- First sub-study: Alcohol-free beer with modified composition (++ maltodextrin) (Experimental): This intervention entails the intake of an alcohol-free beer with modified composition in which the maltose has been almost completely eliminated and enriched with a resistant maltodextrin (2.0 g/100 mL) (MB). This beverage included 25 g of carbohydrates.
  Interventions: Other: Sub-study 1
- Second sub-study: White bread + Water (Active Comparator): This intervention entails the intake of white bread (providing 50 g of carbohydrates) and water.
  Interventions: Other: Sub-study 2
- Second sub-study: White bread + Regular alcohol-free beer (Experimental): This intervention entails the intake of white bread (providing 50 g of carbohydrates) and regular alcohol-free beer (providing 14.3 g of carbohydrates).
  Interventions: Other: Sub-study 2
- Second sub-study: White bread+Alcohol-free beer enriched with isomaltulose+maltodextrin) (Experimental): This intervention entails the intake of white bread (providing 50 g of carbohydrates) and an alcohol-free beer with modified composition in which the maltose has been almost completely eliminated and enriched with isomaltulose (2.5 g/100 mL) and a resistant maltodextrin (0.8 g/100 mL) (IMB). This beverage included 14.3 g of carbohydrates.
  Interventions: Other: Sub-study 2
- Second sub-study: White bread + Alcohol-free beer enriched with ++ maltodextrin (Experimental): This intervention entails the intake of white bread (providing 50 g of carbohydrates) and an alcohol-free beer with modified composition in which the maltose has been almost completely eliminated and enriched a resistant maltodextrin (2.0 g/100 mL) (MB). This beverage included 14.3 g of carbohydrates.
  Interventions: Other: Sub-study 2
- Second sub-study: Extra-White bread + Water (Active Comparator): This intervention entails the intake of white bread which provides 64.3 g (50 g + 14.3 g) of carbohydrates and water. This intervention would be the comparator in carbohydrates-equally conditions.
  Interventions: Other: Sub-study 2

INTERVENTIONS:
Other: Sub-study 1 — Subjects were provided with: a) Glucose beverage; b) Regular alcohol-free beer; c) Alcohol-free beer with modified composition (isomaltulose + maltodextrin); d) Alcohol-free beer with modified composition (++ maltodextrin).
  Arms: First sub-study: Alcohol-free beer with modified composition (++ maltodextrin); First sub-study: Alcohol-free beer with modified composition (isomaltulose + maltodextrin); First sub-study: Glucose beverage; First sub-study: Regular alcohol-free beer
Other: Sub-study 2 — Subjects were provided with: a) White bread + Water; b) White bread + Regular alcohol-free beer; c) White bread+Alcohol-free beer enriched with isomaltulose+maltodextrin); d) White bread + Alcohol-free beer enriched with ++ maltodextrin; e) Extra-White bread + Water.
  Arms: Second sub-study: Extra-White bread + Water; Second sub-study: White bread + Alcohol-free beer enriched with ++ maltodextrin; Second sub-study: White bread + Regular alcohol-free beer; Second sub-study: White bread + Water; Second sub-study: White bread+Alcohol-free beer enriched with isomaltulose+maltodextrin)

SUMMARY:
The overall objective of this study is to explore the glycemic index and glycemic load induced by an alcohol-free beer with modified composition (including almost full fermentation of carbohydrates and the addition of isomaltulose and a resistant maltodextrin), as well as its postprandial metabolic response, compared to the effect induced by: a) an alcohol-free beer with a usual composition; b) an alcohol-free beer with modified composition (including almost full fermentation of carbohydrates and the addition of a resistant maltodextrin). This study includes two cross-over sub-studies recruiting healthy participants. In the first one, 10 healthy volunteers receive 25 g of carbohydrates coming from: regular alcohol-free beer (RB), alcohol-free beer with almost completely eliminated maltose and enriched with isomaltulose (2.5 g/100 mL) and a resistant maltodextrin (0.8 g/100 mL) (IMB), alcohol-free beer with the same maltose removal enriched with resistant maltodextrin (2.0 g/100 mL) (MB) and glucose solution. In the second study, 20 healthy volunteers are provided with 50 g of carbohydrates from white bread and water and the same meal plus 14.3 g of carbohydrates coming from: RB, IMB, MB and extra white bread. Blood is sampled at baseline and for 2 h, every 15 min, after ingestion.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 27.5 kg/m2.

Exclusion Criteria:

* Presence of cardiometabolic pathology such as dyslipemia (total cholesterol > 200 mg/dL and/or triglycerides > 150 mg/dL, and/or taking lipid-lowering drugs), prediabetes or type 1 or 2 diabetes mellitus (glucose ≥ 100 mg/dL and/or glycosylated hemoglobin ≥ 5.7% and/or taking hypoglycemic drugs) or high blood pressure without drug treatment.
* Presence of other chronic pathologies that could interfere with the results of the study such as cardiovascular disease, kidney disease, thyroid disease or liver disease.
* Presence of intestinal malabsorption syndromes and/or presence of Chron disease or ulcerative colitis.
* Use of drugs that may interfere with lipid and/or glycidic metabolism.
* Presence of some analytical alteration that could interfere with the results of the study.
* Increased or decreased body weight of ≥ 5 kg in the last 6 months.
* Gluten intolerance.
* Regular intake of functional foods such as phytosterols or red rice yeast, which have a significant effect on lipid or glycidic metabolism, in the last 6 weeks.
* Intake of vitamin supplements.
* Hormone replacement therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Glucose | Change from Baseline to 15-minutes after consumption of the beverage.
Glucose | Change from Baseline to 30-minutes after consumption of the beverage.
Glucose | Change from Baseline to 45-minutes after consumption of the beverage.
Glucose | Change from Baseline to 60-minutes after consumption of the beverage.
Glucose | Change from Baseline to 75-minutes after consumption of the beverage.
Glucose | Change from Baseline to 90-minutes after consumption of the beverage.
Glucose | Change from Baseline to 105-minutes after consumption of the beverage.
Glucose | Change from Baseline to 120-minutes after consumption of the beverage.
Insulin | Change from Baseline to 15-minutes after consumption of the beverage.
Insulin | Change from Baseline to 30-minutes after consumption of the beverage.
Insulin | Change from Baseline to 45-minutes after consumption of the beverage.
Insulin | Change from Baseline to 60-minutes after consumption of the beverage.
Insulin | Change from Baseline to 75-minutes after consumption of the beverage.
Insulin | Change from Baseline to 90-minutes after consumption of the beverage.
Insulin | Change from Baseline to 105-minutes after consumption of the beverage.
Insulin | Change from Baseline to 120-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 15-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 30-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 45-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 60-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 75-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 90-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 105-minutes after consumption of the beverage.
GLP-1 | Change from Baseline to 120-minutes after consumption of the beverage.
GIP | Change from Baseline to 15-minutes after consumption of the beverage.
GIP | Change from Baseline to 30-minutes after consumption of the beverage.
GIP | Change from Baseline to 45-minutes after consumption of the beverage.
GIP | Change from Baseline to 60-minutes after consumption of the beverage.
GIP | Change from Baseline to 75-minutes after consumption of the beverage.
GIP | Change from Baseline to 90-minutes after consumption of the beverage.
GIP | Change from Baseline to 105-minutes after consumption of the beverage.
GIP | Change from Baseline to 120-minutes after consumption of the beverage.

SECONDARY OUTCOMES:
Leptin | Change from Baseline to 60-minutes after consumption of the beverage.
Leptin | Change from Baseline to 120-minutes after consumption of the beverage.
Glucagon | Change from Baseline to 60-minutes after consumption of the beverage.
Glucagon | Change from Baseline to 120-minutes after consumption of the beverage.
Ghrelin | Change from Baseline to 60-minutes after consumption of the beverage.
Ghrelin | Change from Baseline to 120-minutes after consumption of the beverage.
Polypeptide Y | Change from Baseline to 60-minutes after consumption of the beverage.
Polypeptide Y | Change from Baseline to 120-minutes after consumption of the beverage.
Pancreatic polypeptide | Change from Baseline to 60-minutes after consumption of the beverage.
Pancreatic polypeptide | Change from Baseline to 120-minutes after consumption of the beverage.
HDL cholesterol | Change from Baseline to 60-minutes after consumption of the beverage.
HDL cholesterol | Change from Baseline to 120-minutes after consumption of the beverage.
LDL cholesterol | Change from Baseline to 60-minutes after consumption of the beverage.
LDL cholesterol | Change from Baseline to 120-minutes after consumption of the beverage.
Triglycerides | Change from Baseline to 60-minutes after consumption of the beverage.
Triglycerides | Change from Baseline to 120-minutes after consumption of the beverage.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigación Sanitaria Aragón, Hospital Universitario Miguel Servet, Universidad de Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No